CLINICAL TRIAL: NCT01825837
Title: Extension Study to Investigate the Efficacy, Safety, and Tolerability of Eslicarbazepine Acetate (BIA 2-093) in the Recurrence Prevention of Bipolar I Disorder
Brief Title: Efficacy, Safety, and Tolerability of Eslicarbazepine Acetate in the Recurrence Prevention of Bipolar I Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIA-2093-205
Record Dates: First submitted 2013-04-01; First posted 2013-04-08 (Estimated); Results first posted 2013-06-17 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-02

CONDITIONS: Bipolar I Disorder
Keywords: bipolar I disorder; Eslicarbazepine acetate; BIA 2-093
MeSH Terms: interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- BIA 2-093 1800 mg (Group 1) (Experimental): BIA 2-093 1800 mg once daily (Part II followed a double-blind, parallel-group design in which participants were randomly assigned to treatment with BIA 2-093 300 mg, 900 mg, or 1800 mg once daily). Study medication was administered orally, once daily in the evening.
  Interventions: Drug: BIA 2-093 1800 mg once daily [Group 1 (Part II)]
- BIA 2-093 900 mg (Group 2) (Experimental): BIA 2-093 900 mg once daily (Part II followed a double-blind, parallel-group design in which participants were randomly assigned to treatment with BIA 2-093 300 mg, 900 mg, or 1800 mg once daily). Study medication was administered orally, once daily in the evening.
  Interventions: Drug: BIA 2-093 900 mg once daily [Group 2 (Part II)]
- BIA 2-093 300 mg (Group 3) (Experimental): BIA 2-093 300 mg once daily (Part II followed a double-blind, parallel-group design in which participants were randomly assigned to treatment with BIA 2-093 300 mg, 900 mg, or 1800 mg once daily). Study medication was administered orally, once daily in the evening.
  Interventions: Drug: BIA 2-093 300 mg once daily [Group 3 (Part II)]
- ESL (Part I) (Experimental): In Part I, all participants received open-label treatment with BIA 2-093 900 mg once daily for 2 weeks.
  Interventions: Drug: BIA 2-093 900 mg (Part I)

INTERVENTIONS:
Drug: BIA 2-093 1800 mg once daily [Group 1 (Part II)] — BIA 2-093 1800 mg taken orally in the evening, for 2 weeks
  Other Names: Eslicarbazepine acetate
  Arms: BIA 2-093 1800 mg (Group 1)
Drug: BIA 2-093 900 mg once daily [Group 2 (Part II)] — BIA 2-093 900 mg taken orally in the evening, for 2 weeks
  Other Names: Eslicarbazepine acetate
  Arms: BIA 2-093 900 mg (Group 2)
Drug: BIA 2-093 300 mg once daily [Group 3 (Part II)] — BIA 2-093 300 mg taken orally in the evening, for 2 weeks.
  Other Names: Eslicarbazepine acetate
  Arms: BIA 2-093 300 mg (Group 3)
Drug: BIA 2-093 900 mg (Part I) — In Part I, patients received one 900 mg BIA 2-093 tablet once daily, taken orally in the evening, for 2 weeks.
  Other Names: Eslicarbazepine acetate
  Arms: ESL (Part I)

SUMMARY:
This was an extension study consisting of 2 parts. In Part I, all participants received open-label treatment with BIA 2-093 900 mg once daily for 2 weeks. Part II followed a double-blind, parallel-group design in which participants were randomly assigned to treatment with BIA 2-093 300 mg, 900 mg, or 1800 mg once daily. Patients stable in remission continued double-blind therapy until approximately 6 months after the last patient entered Part II.

DETAILED DESCRIPTION:
The occurrence of a new manic/depressive episode was considered a treatment failure, and the patient was discontinued from the study. At the end of Part II, 6 months after last patient enrolled and after no longer than approximately 15 months, if patients were still in remission and the investigational product was well-tolerated, patients had the option to enter long-term open-label treatment at the same dosage as used in Part II until a new episode occurred, until marketing was authorized, or until clinical development of BIA 2-093 in the recurrence prevention indication was discontinued. If patients did not enter long-term treatment, an established recurrence prevention medication was prescribed, and BIA 2-093 was tapered off (patients assigned to 1800 mg had the daily dose decreased to 900 mg for 6 days; those assigned to 900 mg or 300 mg received placebo for 6 days).

ELIGIBILITY:
Inclusion Criteria:

* signed the Informed consent form (ICF)
* completed the 3-week treatment period in Protocol with identification number SCO/BIA-2093-203 or Protocol with identification number PRA/BIA-2093-204 and shown response to treatment, defined as ≥ 50% improvement in the Young Mania Rating Scale (YMRS) total score or a YMRS total score < 12
* presented a serum pregnancy test (in cases of women of childbearing potential) consistent with a non-gravid state and used double-barrier contraception throughout the study

Exclusion Criteria:

* relevant electrocardiogram (ECG) or laboratory abnormalities
* any uncontrolled clinically relevant disorder
* uninsured capability to comply with the study protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2006-03; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrício Soares-da-Silva, MD, PhD, Study Director — BIAL - Portela & Ca. SA

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study. Approximately 60 centers in Europe, South America, and South Africa enrolled patients in this study.
Pre-assignment Details: This was an extension study consisting of 2 parts. In Part I, all participants received open-label treatment with BIA 2-093 900 mg once daily for 2 weeks. Part II followed a double-blind, parallel-group design in which participants were randomly assigned to treatment with BIA 2-093 300 mg, 900 mg, or 1800 mg once daily
Groups:
- Group 3 [(Part II) 300 mg]: BIA 2-093 300 mg once daily (Part II followed a double-blind, parallel-group design in which participants were randomly assigned to treatment with BIA 2-093 300 mg, 900 mg, or 1800 mg once daily). Study medication was administered orally, once daily in the evening.
- Group 2 [(Part II) 900 mg]: BIA 2-093 900 mg once daily (Part II followed a double-blind, parallel-group design in which participants were randomly assigned to treatment with BIA 2-093 300 mg, 900 mg, or 1800 mg once daily). Study medication was administered orally, once daily in the evening.
- Group 1 [(Part II) 1800 mg]: BIA 2-093 1800 mg once daily (Part II followed a double-blind, parallel-group design in which participants were randomly assigned to treatment with BIA 2-093 300 mg, 900 mg, or 1800 mg once daily). Study medication was administered orally, once daily in the evening.
- ESL (Part I): In Part I, all participants received open-label treatment with BIA 2-093 900 mg once daily for 2 weeks. The participants that completed part I were randomised in Part II.
Period: PART I
Arm/Group | Group 3 [(Part II) 300 mg] | Group 2 [(Part II) 900 mg] | Group 1 [(Part II) 1800 mg] | ESL (Part I)
Started | 0 | 0 | 0 | 104
Enrolled | 0 | 0 | 0 | 104
Safety Population (Open-Label) | 0 | 0 | 0 | 104
Completed | 0 | 0 | 0 | 87
Not Completed | 0 | 0 | 0 | 17
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 6
Not completed — Patient non-compliance | 0 | 0 | 0 | 1
Not completed — Treatment failure | 0 | 0 | 0 | 7
Not completed — reason unspecified | 0 | 0 | 0 | 3
Period: PART II
Arm/Group | Group 3 [(Part II) 300 mg] | Group 2 [(Part II) 900 mg] | Group 1 [(Part II) 1800 mg] | ESL (Part I)
Started | 35 | 26 | 26 | 0
Randomized Patients | 35 | 26 | 26 | 0
Safety Population (Double-Blind) | 35 | 26 | 26 | 0
Intent-to-Treat Population | 34 | 25 | 26 | 0
Per-Protocol Population | 32 | 23 | 24 | 0
Completed | 16 | 12 | 7 | 0
Not Completed | 19 | 14 | 19 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 7 | 0
Not completed — Patient non-compliance | 5 | 2 | 4 | 0
Not completed — Adverse Event | 3 | 3 | 1 | 0
Not completed — Treatment failure | 6 | 4 | 5 | 0
Not completed — reason unspecified | 2 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The study was comprised of 2 sequential parts. Part I followed an open-label design in which all participants received open-label treatment with BIA 2-093 900 mg once daily for 2 weeks. Part II followed a double-blind, parallel-group design in which participants who completed part I. 17 patients did not complete part I.
Groups:
- ESL (Part I - Not Randomised Patients): This group corresponds to the 17 patients who did not complete part I and therefore where not randomised to any traeatment group.
- Total: Total of all reporting groups
Arm/Group | Group 3 [(Part II) 300 mg] | Group 2 [(Part II) 900 mg] | Group 1 [(Part II) 1800 mg] | ESL (Part I - Not Randomised Patients) | Total
Number analyzed (Participants) | 35 | 26 | 26 | 17 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 24 | 25 | 17 | 100
  >=65 years | 1 | 2 | 1 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 11 | 12 | 50
  Male | 19 | 15 | 15 | 5 | 54

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Showed no Worsening According to the Clinical Global Impression - Bipolar Version (CGI-BP) Scale (Intent-to-Treat Population)
Description: The CGI-BP scale is a modification of the CGI scale, which provides a means of assessing severity and treatment-related improvement in manic and depressive domains reflecting clinically relevant degrees of change. The concept of improvement refers to the clinical distance between the individual's current condition and that prior to the start of treatment. The scale for 'severity of illness' measures mania, depression and overall illness on a 7 point scale from 1 ('normal, not ill') to 7 ('very severely ill'). The scale for 'change from preceding phase' and 'change from worst phase' measures mania, depression, and overall illness on an 8-point scale from 1 (very much improved) to 8 ('not applicable'). If the patient, in 'change from preceding phase', at any visit during the double-blind, has a score of 5, 6, or 7 in any of 3 categories (mania, depression, or overall bipolar illness), then the illness will be considered to have worsened.
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- BIA 2-093 300 mg; BIA 2-093 900 mg; BIA 2-093 1800 mg: PART II - Intent-to-Treat Population
Arm/Group | BIA 2-093 300 mg | BIA 2-093 900 mg | BIA 2-093 1800 mg
Number analyzed (Participants) | 34 | 25 | 26
participants | 26 | 14 | 16

ADVERSE EVENTS:
Time Frame: Double-blind period (Part II first administration date until study termination) 6 months
Description: Part II Double-Blind Period (Safety Population): safety population included all patients who received at least 1 dose of investigational product after randomization. Please note that adverse events that occurred in Parts I and II were summarized separately.
Arm/Group | Group 3 [(Part II) 300 mg] | Group 2 [(Part II) 900 mg] | Group 1 [(Part II) 1800 mg]
Serious Adverse Events (participants affected / at risk) | 2/35 | 4/26 | 2/26
Other Adverse Events (participants affected / at risk) | 7/35 | 6/26 | 4/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 3 [(Part II) 300 mg] (N=35) | Group 2 [(Part II) 900 mg] (N=26) | Group 1 [(Part II) 1800 mg] (N=26)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 3 [(Part II) 300 mg] (N=35) | Group 2 [(Part II) 900 mg] (N=26) | Group 1 [(Part II) 1800 mg] (N=26)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (1) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood pressure systolic decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other